CLINICAL TRIAL: NCT04416412
Title: Optimizing Surgical Debridement Following High-energy Open Trauma With Dynamic Contrast-enhanced Fluorescence Imaging
Brief Title: ICG Fluorescence Imaging in Open Fracture Trauma Patients
Status: Active, not recruiting | Type: Observational
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Dartmouth College (Other); United States Department of Defense (U.S. Federal Agency); Brigham and Women's Hospital (Other); University of California, Irvine (Other); University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Ida Leah Gitajn, Physician, Dartmouth-Hitchcock Medical Center
Other Study IDs: D20058; OR190062 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2020-05-21; First posted 2020-06-04 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-03

CONDITIONS: Trauma Injury
Keywords: Immunofluorescence; Orthopaedic; Trauma; Open Fracture
MeSH Terms: conditions — Accidental Injuries; Wounds and Injuries; Fractures, Open

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Open Fracture Cohort: Patients 18 years of age or older. Open extremity fracture. Planned definitive fracture management with external fixation, internal fixation, or joint fusion.
  Open fracture wound management that includes formal surgical debridement within 72 hours of their injury.
  Will have all planned fracture care surgeries performed by a participating surgeon or delegate.
  Provision of informed consent.
  Interventions: Other: Immunofluorescence Imaging

INTERVENTIONS:
Other: Immunofluorescence Imaging — Patients will be administered FDA approved ICG through intravenous injection and imaged by a FDA approved surgical microscope (Spy Elite) which is 0.5 meter away from the subject. Both ICG fluorescence and the two imaging systems have been used for routine clinical practice for many years. Figure (a) shows the Schematic sketch of the imaging systems. ICG fluorescence imaging utilizes intravenously injected ICG, which is a fluorescent dye that is FDA-approved for clinical use, illuminated with near-infrared light. The ICG dye is indirectly activated and the dynamic fluorescence due to bone perfusion can be captured by a video rate imaging system.

SUMMARY:
This is a prospective observational study that will evaluate the association between bone and tissue perfusion, as measured by indocyanine green (ICG) fluorescence imaging, and complications, in an effort to develop ICG fluorescence imaging as a diagnostic tool to quantitatively guide operative debridement.

DETAILED DESCRIPTION:
This is a prospective observational study that will evaluate the association between bone and tissue perfusion, as measured using indocyanine green (ICG) fluorescence imaging, and complications. This will be used to develop ICG fluorescence imaging as a diagnostic tool to objectively and quantitatively guide operative debridement. The study population includes all open fracture patients regardless of race, ethnicity, or sex/gender. Primary outcome measure is all-cause re-operation and secondary outcome measure is surgical site infection. All patients will be followed for a total of 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 years of age or older.
2. Open extremity fracture.
3. Planned definitive fracture management with external fixation, internal fixation, or joint fusion.
4. Open fracture wound management that includes formal surgical debridement within 72 hours of their injury.
5. Will have all planned fracture care surgeries performed by a participating surgeon or delegate.
6. Provision of informed consent.

Exclusion Criteria:

1. Inability of patient to provide informed consent
2. Fracture of the hand.
3. Iodine allergy.
4. Received previous surgical debridement or management of their fracture at a non-participating hospital or clinic.
5. Open fracture managed outside of the participating orthopaedic service.
6. Chronic or acute infection at or near the fracture site at the time of initial fracture surgery.
7. Burns at the fracture site.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 18 years of age or older who present with an open fracture will be considered for the open fracture cohort.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants who undergo an unplanned fracture-related reoperation | 12 months
  All unplanned reoperations will be documented using a specific case report form
Number of participants who experience a post-procedure surgical site infection | 12 months
  Post-procedure surgical site infection using Centers for Disease Control criteria will be documented at each follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Ida L Gitajn, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (4):
- United States (4):
  - University of California, Irvine, Irvine, California
  - University of Maryland, Baltimore R. Cowley Shock Trauma, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire

IPD SHARING:
Plan to Share IPD: No